CLINICAL TRIAL: NCT06366321
Title: Using Digital Technology Versus Conventional Relining Procedure for Correction of Loose Maxillary Complete Denture. Crossover Randomized Control Trial.
Brief Title: Using Digital Technology Versus Conventional Relining Procedure for Correction of Loose Maxillary Complete Denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Maha kamal, Associate professor, British University In Egypt
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 23-067
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Dental Diseases; Dental Trauma; Bone Remodeling Disorder
Keywords: Relining upper denture; Digital denture; Denture Retention; Denture adaptation.; CAD/CAM milling
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventionally constructed denture (Other): construction of complete dentures by conventional (lost wax casting) technique
  Interventions: Other: relining technique
- digitally constructed denture (Other): construction of complete dentures by digital (CAD/CAM milling) technique
  Interventions: Other: CAD/CAM milling technique

INTERVENTIONS:
Other: relining technique — construction of complete denture by flasking and casting the relining impression
  Other Names: no other names
  Arms: conventionally constructed denture
Other: CAD/CAM milling technique — construction of complete denture by milling of the scanned relining impression
  Other Names: computer added designing/ computer added milling
  Arms: digitally constructed denture

SUMMARY:
This study aimed to evaluate the use of computer added designning / computer added manufacturing (CAD/ CAM ) technology versus conventional relining procedure for treating ill-fitted loose maxillary complete denture and its effect on patient satisfaction, denture retention, and denture adaptation to oral tissues.

DETAILED DESCRIPTION:
Twelve edentulous patients suffering from loose maxillary complete dentures were selected, the dentures were adjusted for taking the relining impressions, the impressions were scanned and the STL files were used for milling new dentures (Group A), then the relining impression went through the conventional laboratory steps of processing (Group B). Both groups were evaluated regarding patient's satisfaction by a specially designed questionnaire, retention values were measured by a digital force gauge at denture insertion appointment and two weeks later, finally dentures adaptation to the oral tissues were compared using geomagic software.

ELIGIBILITY:
Inclusion Criteria:

* Patients with completely edentulous maxillary and mandibular ridges with a normal skeletal relationship (class I) have a moderate-to-highly well-rounded maxillary edentulous ridge without severe undercuts to minimize the effect of undercuts on retention values.
* Patients' main complaint was a loose or "falling" denture, but with proper esthetics, centric relation and the correct vertical dimension of occlusion (VDO).

Exclusion Criteria:

* Patients with significant skeletal problems (class II or III) or who went through severe osseous surgery or any hereditary or acquired osseous abnormality find it challenging to place the denture properly on the supporting ridge.
* If the patient suffers from xerostomia, excessive flabby ridges, any pathology of the oral mucosa, or any inflammatory changes, candidiasis, hyperplasia, neurological disorders and malignancies
* If the denture creates a major speech problem, poor esthetics, or an unsatisfactory jaw relationship.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
patient satisfaction using questionnaire | two week
  A version of Likert scale with ranges from 1 (completely unsatisfied) to 5 (completely satisfied) was used representing the denture satisfaction scale at denture insertion time and two weeks later regarding denture retention, improved mastication, proper speech, and esthetics.
  Patient-based outcomes data were collected. A total satisfaction score was calculated of each item; higher scores mean greater satisfaction.
denture retention | two weeks
  * An (19-gauge) orthodontic wire in the form of a hook was secured on the center of the palate at a point of intersection of the lines connecting the hamular notches, the right and left canines with the midline by self-cured acrylic resin material and placed on the supporting tissues intraorally.
  * Testing procedure: The patient was in an upright position. Digital force gauge (Force Gauge HF- 50N) was linked to the hook and a downward pulled force was applied slowly in a vertical direction opposite to that of the denture path of insertion until the denture was displaced and the highest force value was registered. After completing this procedure three times, the average was determined.
denture adaptation to oral tissues | at the time of denture insertion
  * Maxillary arches of all patients were scanned using intraoral scanner (3 shape TRIOS 4 wired, Copenhagen, Denmark), fitting surfaces of both denture groups were also scanned using desktop scanner ( 3Shape E2, Copenhagen, Denmark) then A 3D measurement program (Geomagic Control X, 3D Systems, United States) was used to build and superimpose STL files using first initial alignment and then best-fit alignment (fig 7 A&B). For every measurement point, the root mean square (RMS) (mm) was computed considering both positive and negative values.
  * Color map of CAD/CAM milled denture's fitting surface adaptation and of conventionally relined denture's fitting surface adaptation was formed, pressure from the denture fitting surface to the oral tissues is indicated by yellow to red colors. The denture fitting surface and oral tissues are separated by a blue color. Green color denotes that the oral tissues and the denture fitting surface are in contact.

CONTACTS AND LOCATIONS:
Overall Officials: maha kamal, A. Professor, Principal Investigator — British University In Egypt
Locations (1):
- British University in Egypt, El Shorouk, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamal MNM. Comparison between relining of ill-fitted maxillary complete denture versus CAD/CAM milling of new one regarding patient satisfaction, denture retention and adaptation. BMC Oral Health. 2025 Jan 4;25(1):18. doi: 10.1186/s12903-024-05298-z. PMID 39755611